CLINICAL TRIAL: NCT03934385
Title: Optimizing Exposure Therapy With Mental Rehearsal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Anastasia McGlade, MA, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AM74RL539
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Anxiety Disorders; Arachnophobia
Keywords: anxiety; consolidation; extinction; mental rehearsal
MeSH Terms: conditions — Anxiety Disorders; Arachnophobia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Rehearsal (Experimental): Between-session rehearsal/retrieval exercises focused upon consolidating non-fear learning gained from exposures by prompting reflection of expectancy violation and rehearsal of the inhibitory association between the conditioned stimulus (i.e., spider) and unconditioned stimulus (e.g., bite/attack).
  Interventions: Behavioral: Mental Rehearsal; Behavioral: Exposure
- Control Rehearsal (Active Comparator): Between-session rehearsal/retrieval exercises focused upon an unrelated, recent academic experience.
  Interventions: Behavioral: Exposure

INTERVENTIONS:
Behavioral: Mental Rehearsal — After each exposure session, participants complete three rehearsal/retrieval exercises that involve viewing images of spiders and completing multiple-choice and free-response questions. Exercises involve retrieving information specific to the spider exposures, reflecting on the experience, and highlighting expectancy violation (i.e., that the participant's feared outcome did not occur).
  Other Names: mental retrieval
  Arms: Mental Rehearsal
Behavioral: Exposure — All participants complete two exposure sessions. The first set of exposures consists of ten 30-second trials hovering one's hand 3 inches over a live tarantula. The second set of exposures consists of ten 30-second trials placing one's hand inside the spider's terrarium with all five fingertips touching the bottom.

SUMMARY:
Treatment response rates for cognitive behavioral therapy (CBT) across anxiety disorders average approximately 50% post-treatment (Loerinc et al, 2015), evidencing significant 'return of fear', the re-emergence of a partially or fully extinguished fear (Rachman, 1989). Thus, recent research has amplified efforts toward improving treatment methodology in an attempt to optimize clinical outcomes. Many efforts have targeted exposure therapy, an evidence-based behavioral technique during which a patient is strategically and repeatedly exposed to his or her feared stimulus in an effort to generate new non-fear associations with that stimulus. One such effort involves mental rehearsal, where information is reinstated using either a cue from extinction training or imaginal recounting of previous successful exposures (Craske et al, 2014). Prior research has assessed the effects of mental rehearsal via reinstatement of the extinction context (i.e., treatment context) or of cues/items from the treatment context that may indicate safety (e.g., Mystkowski et al, 2006; Culver, Stoyanova, & Craske, 2011). However, this research has produced inconsistent results and contains an inherent limitation, as retrieval cues may become a safety signal and inhibit new learning (Dibbets, Havermans, & Arntz, 2008).

In an effort to address these limitations, the current study recruits spider-fearful participants for a treatment trial consisting of exposures in conjunction with either a mental rehearsal intervention, or a control rehearsal intervention. The overarching goal of this project is to evaluate the extent to which a between-session, technology-guided mental rehearsal intervention may optimize exposure therapy outcomes. We also seek to evaluate potential mechanisms of mental rehearsal.

Participants complete three laboratory visits, including two sessions of exposures with live spiders. Participants are randomized to either a mental rehearsal or control rehearsal condition to measure potential mechanisms and moderators of mental rehearsal. Laboratory-based assessments include measures of subjective, behavioral, and psychophysiological responses to spiders.

DETAILED DESCRIPTION:
Return of fear is the re-emergence of a partially or fully extinguished fear (Rachman, 1989). Due to relatively low treatment response rates for CBT at post-treatment (Loerinc et al, 2015), this study seeks to assess the efficacy of mental rehearsal (MR) in a different, less context-dependent manner than prior efforts (e.g., Mystkowski et al, 2006; Culver, Stoyanova, & Craske, 2011). Participants in the MR condition rehearse the new learning contingency, that is, that their feared outcome did not occur when they approached a live spider. Violation of expectancies engenders new, secondary learning that competes with the older fear memory (Craske et al, 2008; Bjork, 2003). As secondary, non-fear learning is repeatedly retrieved, the original fear memory is gradually suppressed, rendering it less recallable in the future (Bjork, 2011). Thus, repeatedly retrieving non-fear learning acquired from exposures is purported to strengthen the non-fear memory and reduce symptoms of arachnophobia. MR is conducted between sessions in an effort to reduce short-term return of fear by enhancing consolidation of non-fear learning via rehearsal efforts in multiple environments/contexts.

The overall aim of the current study is to evaluate a method for enhancing the effectiveness of exposure therapy, and more specifically, to test the extent to which a novel between-session mental rehearsal intervention may optimize treatment outcomes in individuals with excessive fear of spiders. An important secondary aim is to better understand cognitive and affective mechanisms underlying benefits of mental rehearsal.

The experiment consists of three sessions, spanning 8-10 days. Session 1 begins with a pre-treatment assessment consisting of self-report questionnaires and a behavioral approach test (BAT) with a live spider. During the BAT, confidence and distress ratings are obtained and psychophysiological responses (i.e., SCR) are recorded. Participants then complete a series of exposures with a live spider. At Session 2 (two to three days later), participants return to complete a second series of exposures with a live spider. At Session 3 (five to seven days later), participants complete a post-treatment assessment with self-report questionnaires and BAT, again with concurrent confidence and distress ratings and psychophysiological recordings.

Between sessions, participants are randomized to mentally rehearse information from exposures (i.e., MR) or from an unrelated recent academic experience (i.e., Control). MR exercises guide participants in retrieving and consolidating learning from exposures, emphasizing the inhibitory relationship between the conditioned stimulus (CS) and the unconditioned stimulus (US) (i.e., that approaching the spider did not result in their anticipated/feared outcome).

Measures span self-report, behavioral, and psychophysiological data. Fear of spiders is assessed with self-reported symptoms and measures taken during pre- and post-treatment BATs. During each BAT, skin conductance response (SCR) serves as a physiological index of fearful arousal. Baseline SCR is collected during a two-minute period at the start of pre- and post-treatment assessments. At both BATs, anticipatory SCR is collected during a one-minute period immediately prior to starting the BAT, and SCR is then continuously recorded throughout completion of the BAT. In addition to SCR, number of steps completed (0 to 9) and repeated ratings of confidence, anticipatory distress, and maximum distress during the BAT serve as important indices of fear.

Self-reported stress, sleep quality, aerobic exercise, and knowledge of spiders are assessed as potential moderators of mental rehearsal and symptom change. Post-exposure ratings of surprise, US expectancy, and generalization of non-fear learning will additionally be evaluated as treatment mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Elevated score on Spider Phobia Questionnaire (SPQ)

Exclusion Criteria:

* Severe allergies to bees/spiders/insects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Spider Phobia Questionnaire (SPQ; Klorman et al, 1974) | Change from baseline to post-treatment (i.e., 8-10 days)
  31-item true/false questionnaire assessing symptoms of arachnophobia. Scores range from 0 to 31, with greater scores representing greater fear of spiders. Spider phobic individuals have obtained mean scores of 23.20 (SD = 2.90) and 23.76 (SD = 3.80) on the SPQ (Klorman et al, 1974; Murris & Merckelbach, 1996).
Behavioral Approach Test (BAT) steps | Change from baseline to post-treatment (i.e., 8-10 days)
  Number of test steps fully completed
SCR anticipation | Change from baseline to post-treatment (i.e., 8-10 days)
  Change in SCR from baseline to BAT anticipation
SCR across BAT steps | Change from baseline to post-treatment (i.e., 8-10 days)
  SCR during each 30-second test step fully completed
Confidence ratings | Change from baseline to post-treatment (i.e., 8-10 days)
  Repeated confidence ratings on a scale from 0 (no confidence) to 100 (complete confidence) recorded throughout BAT
Distress ratings | Change from baseline to post-treatment (i.e., 8-10 days)
  Repeated anticipatory and maximum distress ratings on a scale from 0 (no distress) to 100 (severe distress) recorded throughout BAT

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales (DASS-21; Lovibond & Lovibond, 1995) | Baseline
  21-item self-report measure that assesses severity of symptoms of depression, anxiety, and stress. We use scores on the Stress subscale, which consists of 7 items measuring chronic non-specific arousal (e.g., difficulty relaxing, nervous energy, agitation, irritability). The minimum score on this subscale is 0 and the maximum score is 42 (0-14 = normal, 15-18 = mild, 19-25 = moderate, 26-33 = severe, 34+ = extremely severe).
Pittsburgh Sleep Quality Index (PSQI; Buysse et al, 1989) | Baseline
  18-item self-report measure that assesses sleep quality and disturbances over the past month. We use the global score, which sums seven component scores. Scores range from 0 to 21, with a score of 5 or greater indicating poor sleep quality.
Aerobic exercise | Baseline
  Brief 4-item self-report measure that assesses time spent doing scheduled and unscheduled aerobic activity during a typical week.
Surprise | Session 1 and Session 2 (i.e., 3 days)
  Ratings of surprise on a 5-pt Likert scale (1 = not at all surprised, 5 = extremely surprised) concerning the outcome of exposures. Scores are averaged across two exposure sessions. Scores range from 1 to 5, with greater values indicating greater surprise with the outcome of exposures.
US expectancy | Session 1 and Session 2 (i.e., 3 days)
  Ratings of US expectancy on a 5-pt Likert scale (0 = not at all likely, 5 = extremely likely) concerning a participant's estimated likelihood of the feared outcome occurring with the same context and stimulus as in vivo exposures. Scores are averaged across two exposure sessions. Scores range from 1 to 5, with greater values indicating greater US expectancy post-exposures.
Non-fear generalization | Session 1 and Session 2 (i.e., 3 days)
  Ratings of US expectancy on a 5-pt Likert scale (0 = not at all likely, 5 = extremely likely) concerning a participant's estimated likelihood of the feared outcome occurring with a different spider outside the lab. Scores are averaged across two exposure sessions. Scores range from 1 to 5, with lower values indicating greater ability to generalize safety learning.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia L McGlade, MA, Principal Investigator — University of California, Los Angeles; Michelle G Craske, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Anderson MC, Bjork RA, Bjork EL. Remembering can cause forgetting: retrieval dynamics in long-term memory. J Exp Psychol Learn Mem Cogn. 1994 Sep;20(5):1063-87. doi: 10.1037//0278-7393.20.5.1063. PMID 7931095
- [Background] Aubry AV, Serrano PA, Burghardt NS. Molecular Mechanisms of Stress-Induced Increases in Fear Memory Consolidation within the Amygdala. Front Behav Neurosci. 2016 Oct 21;10:191. doi: 10.3389/fnbeh.2016.00191. eCollection 2016. PMID 27818625
- [Background] Bjork, E. L., & Bjork, R. A. (2011). Making things hard on yourself, but in a good way: Creating desirable difficulties to enhance learning. In M. A. Gernsbacher, R. W. Pew, L. M. Hough, J. R. Pomerantz (Eds.) & FABBS Foundation, Psychology and the real world: Essays illustrating fundamental contributions to society (pp. 56-64). New York, NY, US: Worth Publishers.
- [Background] Bjork, R. A. (2003). Interference and forgetting. In J. H. Byrne (Ed.), Encyclopedia of learning and memory, 2nd ed., (pp. 268-273). New York: Macmillan Reference USA.
- [Background] Bjork, R.A. (2011). On the symbiosis of learning, remembering, and forgetting. In A. S. Benjamin (Ed.), Successful remembering and successful forgetting: a Festschrift in honor of Robert A. Bjork (pp. 1-22). London, UK: Psychology Press.
- [Background] Bjork, R. A., & Bjork, E. L. (1992). A new theory of disuse and an old theory of stimulus fluctuation. In A. Healy, S. Kosslyn, & R. Shiffrin (Eds.), From learning processes to cognitive processes: Essays in honor of William K. Estes (pp. 35-67). Hillsdale, NJ: Erlbaum.
- [Background] Bloom, K. C., & Shuell, T. J. (1981). Effects of massed and distributed practice on the learning and retention of second-language vocabulary. The Journal of Educational Research, 74(4), 245-248. doi:10.1080/00220671.1981.10885317
- [Background] Bouton, M. E., & Swartzentruber, D. (1991). Sources of relapse after extinction in Pavlovian and instrumental learning. Clinical Psychology Review, 11, 123-140. doi:10.1016/0272-7358(91)90091-8
- [Background] Bouton ME, Westbrook RF, Corcoran KA, Maren S. Contextual and temporal modulation of extinction: behavioral and biological mechanisms. Biol Psychiatry. 2006 Aug 15;60(4):352-60. doi: 10.1016/j.biopsych.2005.12.015. Epub 2006 Apr 17. PMID 16616731
- [Background] Bramham CR, Messaoudi E. BDNF function in adult synaptic plasticity: the synaptic consolidation hypothesis. Prog Neurobiol. 2005 Jun;76(2):99-125. doi: 10.1016/j.pneurobio.2005.06.003. PMID 16099088
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cahill L, Gorski L, Le K. Enhanced human memory consolidation with post-learning stress: interaction with the degree of arousal at encoding. Learn Mem. 2003 Jul-Aug;10(4):270-4. doi: 10.1101/lm.62403. PMID 12888545
- [Background] Cahill L, McGaugh JL. A novel demonstration of enhanced memory associated with emotional arousal. Conscious Cogn. 1995 Dec;4(4):410-21. doi: 10.1006/ccog.1995.1048. PMID 8750416
- [Background] Cain CK, Blouin AM, Barad M. Adrenergic transmission facilitates extinction of conditional fear in mice. Learn Mem. 2004 Mar-Apr;11(2):179-87. doi: 10.1101/lm.71504. PMID 15054133
- [Background] Choy Y, Fyer AJ, Lipsitz JD. Treatment of specific phobia in adults. Clin Psychol Rev. 2007 Apr;27(3):266-86. doi: 10.1016/j.cpr.2006.10.002. Epub 2006 Nov 15. PMID 17112646
- [Background] Christopoulos, G. I., Uy, M. A., & Yap, W. J. (2016). The body and the brain: measuring skin conductance response to understand the emotional experience. Organizational Research Methods, 1-27. doi:10.1177/1094428116681073
- [Background] Cotman CW, Berchtold NC, Christie LA. Exercise builds brain health: key roles of growth factor cascades and inflammation. Trends Neurosci. 2007 Sep;30(9):464-72. doi: 10.1016/j.tins.2007.06.011. Epub 2007 Aug 31. PMID 17765329
- [Background] Craske MG, Kircanski K, Zelikowsky M, Mystkowski J, Chowdhury N, Baker A. Optimizing inhibitory learning during exposure therapy. Behav Res Ther. 2008 Jan;46(1):5-27. doi: 10.1016/j.brat.2007.10.003. Epub 2007 Oct 7. PMID 18005936
- [Background] Craske MG, Treanor M, Conway CC, Zbozinek T, Vervliet B. Maximizing exposure therapy: an inhibitory learning approach. Behav Res Ther. 2014 Jul;58:10-23. doi: 10.1016/j.brat.2014.04.006. Epub 2014 May 9. PMID 24864005
- [Background] Culver NC, Stoyanova M, Craske MG. Clinical relevance of retrieval cues for attenuating context renewal of fear. J Anxiety Disord. 2011 Mar;25(2):284-92. doi: 10.1016/j.janxdis.2010.10.002. Epub 2010 Nov 3. PMID 21146358
- [Background] Dibbets P, Havermans R, Arntz A. All we need is a cue to remember: the effect of an extinction cue on renewal. Behav Res Ther. 2008 Sep;46(9):1070-7. doi: 10.1016/j.brat.2008.05.007. Epub 2008 Jun 27. PMID 18675398
- [Background] Donovan, J. J., & Radosevich, D. J. (1999). A meta-analytic review of the distribution of practice effect: Now you see it, now you don't. Journal of Applied Psychology, 84(5), 795-805. doi:10.1037/0021-9010.84.5.795
- [Background] Driskell, J. E., Willis, R. P., & Copper, C. (1992). Effect of overlearning on retention. Journal of Applied Psychology, 77, 615-622. doi:10.1037/0021-9010.77.5.615
- [Background] Dunsmoor JE, Paz R. Fear Generalization and Anxiety: Behavioral and Neural Mechanisms. Biol Psychiatry. 2015 Sep 1;78(5):336-43. doi: 10.1016/j.biopsych.2015.04.010. Epub 2015 Apr 20. PMID 25981173
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Hofmann SG, Smits JA. Cognitive-behavioral therapy for adult anxiety disorders: a meta-analysis of randomized placebo-controlled trials. J Clin Psychiatry. 2008 Apr;69(4):621-32. doi: 10.4088/jcp.v69n0415. PMID 18363421
- [Background] Hotting K, Schickert N, Kaiser J, Roder B, Schmidt-Kassow M. The Effects of Acute Physical Exercise on Memory, Peripheral BDNF, and Cortisol in Young Adults. Neural Plast. 2016;2016:6860573. doi: 10.1155/2016/6860573. Epub 2016 Jun 29. PMID 27437149
- [Background] Kalueff AV. Neurobiology of memory and anxiety: from genes to behavior. Neural Plast. 2007;2007:78171. doi: 10.1155/2007/78171. Epub 2007 Jan 10. PMID 17502911
- [Background] Karpicke JD, Roediger HL 3rd. The critical importance of retrieval for learning. Science. 2008 Feb 15;319(5865):966-8. doi: 10.1126/science.1152408. PMID 18276894
- [Background] Kircanski K, Lieberman MD, Craske MG. Feelings into words: contributions of language to exposure therapy. Psychol Sci. 2012 Oct 1;23(10):1086-91. doi: 10.1177/0956797612443830. Epub 2012 Aug 16. PMID 22902568
- [Background] Klorman, R., Weerts, T.C., Hastings, J.E., Melamed, B.G., Lang, P.J. (1974). Psychometric descriptions of some specific fear questionnaires. Behavior Therapy, 5, 401-409. doi:10.1016/S0005-7894(74)80008-0
- [Background] Laine CM, Spitler KM, Mosher CP, Gothard KM. Behavioral triggers of skin conductance responses and their neural correlates in the primate amygdala. J Neurophysiol. 2009 Apr;101(4):1749-54. doi: 10.1152/jn.91110.2008. Epub 2009 Jan 14. PMID 19144740
- [Background] Lang AJ, Craske MG. Manipulations of exposure-based therapy to reduce return of fear: a replication. Behav Res Ther. 2000 Jan;38(1):1-12. doi: 10.1016/s0005-7967(99)00031-5. PMID 10645020
- [Background] Lang, A. J., Craske, M. G., & Bjork, R. A. (1999). Implications of a new theory of disuse for the treatment of emotional disorders. Clinical Psychology: Science and Practice, 6, 80-94. doi:10.1093/clipsy/6.1.80
- [Background] Litman L, Davachi L. Distributed learning enhances relational memory consolidation. Learn Mem. 2008 Aug 26;15(9):711-6. doi: 10.1101/lm.1132008. Print 2008 Sep. PMID 18772260
- [Background] Loerinc AG, Meuret AE, Twohig MP, Rosenfield D, Bluett EJ, Craske MG. Response rates for CBT for anxiety disorders: Need for standardized criteria. Clin Psychol Rev. 2015 Dec;42:72-82. doi: 10.1016/j.cpr.2015.08.004. Epub 2015 Aug 14. PMID 26319194
- [Background] Lovibond, S.H. & Lovibond, P.F. (1995). Manual for the Depression Anxiety Stress Scales. (2nd Ed.) Sydney: Psychology Foundation.
- [Background] McGaugh JL. Consolidating memories. Annu Rev Psychol. 2015 Jan 3;66:1-24. doi: 10.1146/annurev-psych-010814-014954. PMID 25559113
- [Background] Meeter M, Murre JM. Consolidation of long-term memory: evidence and alternatives. Psychol Bull. 2004 Nov;130(6):843-57. doi: 10.1037/0033-2909.130.6.843. PMID 15535740
- [Background] Meuret AE, Rosenfield D, Bhaskara L, Auchus R, Liberzon I, Ritz T, Abelson JL. Timing matters: Endogenous cortisol mediates benefits from early-day psychotherapy. Psychoneuroendocrinology. 2016 Dec;74:197-202. doi: 10.1016/j.psyneuen.2016.09.008. Epub 2016 Sep 15. PMID 27664810
- [Background] Meuret AE, Trueba AF, Abelson JL, Liberzon I, Auchus R, Bhaskara L, Ritz T, Rosenfield D. High cortisol awakening response and cortisol levels moderate exposure-based psychotherapy success. Psychoneuroendocrinology. 2015 Jan;51:331-40. doi: 10.1016/j.psyneuen.2014.10.008. Epub 2014 Oct 16. PMID 25462905
- [Background] Muris P, Merckelbach H. A comparison of two spider fear questionnaires. J Behav Ther Exp Psychiatry. 1996 Sep;27(3):241-4. doi: 10.1016/s0005-7916(96)00022-5. PMID 8959425
- [Background] Mystkowski JL, Craske MG, Echiverri AM, Labus JS. Mental reinstatement of context and return of fear in spider-fearful participants. Behav Ther. 2006 Mar;37(1):49-60. doi: 10.1016/j.beth.2005.04.001. Epub 2006 Feb 24. PMID 16942960
- [Background] Rachman, S. (1989). The return of fear: Review and prospect. Clinical Psychology Review, 9, 147-168. doi:10.1016/0272-7358(89)90025-1
- [Background] Rasch B, Born J. About sleep's role in memory. Physiol Rev. 2013 Apr;93(2):681-766. doi: 10.1152/physrev.00032.2012. PMID 23589831
- [Background] Rodriguez BI, Craske MG, Mineka S, Hladek D. Context-specificity of relapse: effects of therapist and environmental context on return of fear. Behav Res Ther. 1999 Sep;37(9):845-62. doi: 10.1016/s0005-7967(98)00106-5. PMID 10458048
- [Background] Rowe MK, Craske MG. Effects of an expanding-spaced vs massed exposure schedule on fear reduction and return of fear. Behav Res Ther. 1998 Jul-Aug;36(7-8):701-17. doi: 10.1016/s0005-7967(97)10016-x. PMID 9682526
- [Background] Rowe MK, Craske MG. Effects of varied-stimulus exposure training on fear reduction and return of fear. Behav Res Ther. 1998 Jul-Aug;36(7-8):719-34. doi: 10.1016/s0005-7967(97)10017-1. PMID 9682527
- [Background] Soule J, Messaoudi E, Bramham CR. Brain-derived neurotrophic factor and control of synaptic consolidation in the adult brain. Biochem Soc Trans. 2006 Aug;34(Pt 4):600-4. doi: 10.1042/BST0340600. PMID 16856871
- [Background] Squire LR. Memory and the hippocampus: a synthesis from findings with rats, monkeys, and humans. Psychol Rev. 1992 Apr;99(2):195-231. doi: 10.1037/0033-295x.99.2.195. PMID 1594723
- [Background] Vervliet B, Craske MG, Hermans D. Fear extinction and relapse: state of the art. Annu Rev Clin Psychol. 2013;9:215-48. doi: 10.1146/annurev-clinpsy-050212-185542. PMID 23537484
- [Background] Wolitzky-Taylor KB, Horowitz JD, Powers MB, Telch MJ. Psychological approaches in the treatment of specific phobias: a meta-analysis. Clin Psychol Rev. 2008 Jul;28(6):1021-37. doi: 10.1016/j.cpr.2008.02.007. Epub 2008 Mar 7. PMID 18410984